CLINICAL TRIAL: NCT06196723
Title: TIPS Improve Survival in Patients With Cirrhosis and Recurrent Ascites: a Multicenter Observational Study
Brief Title: Transjugular Intrahepatic Portosystemic Shunts Improve Survival in Patients With Cirrhosis and Recurrent Ascites
Acronym: TIPS
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Xijing Hospital
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Refractory Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TIPS: transjugular intrahepatic portal shunt
  Interventions: Procedure: transjugular intrahepatic portal shunt
- LVP+A: large volume paracenteses plus albumin

INTERVENTIONS:
Procedure: transjugular intrahepatic portal shunt — TIPS was performed by experienced clinicians in the Gastroenterology/Hepatology Department according to standard operating procedures, utilizing 8 mm or 10 mm expanded polytetrafluoroethylene-covered stents at the discretion of the local physician.
  Groups: TIPS

SUMMARY:
Currently, there is limited evidence regarding the survival benefit of early transjugular intrahepatic portal shunt (TIPS) placement in patients with cirrhosis and recurrent ascites. This observational study aimed to assess whether early TIPS improves the survival of patients with advanced cirrhosis and recurrent ascites. We will compare large volume paracenteses plus albumin (LVP+A） to see if TIPS improves the survival of patients with advanced cirrhosis and recurrent ascites.

ELIGIBILITY:
Inclusion Criteria:

Definite diagnosis of recurrent ascites in cirrhosis (based on clinical symptoms, laboratory and imaging studies, or liver biopsy) TIPS or LVP+A therapy, -

Exclusion Criteria:

Malignant neoplasm, including hepatocellular carcinoma with extrahepatic metastasis Prior liver transplantation Severe heart and lung dysfunction Recurrent hepatic encephalopathy Concomitant active infection TIPS with the use of uncovered stents Complete portal vein thrombosis

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included patients with cirrhosis and recurrent ascites who were treated with TIPS or large volume paracenteses plus albumin at 11 tertiary level A hospitals in China
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
One year transplant free survival | One year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Tangdu hospital, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No